CLINICAL TRIAL: NCT01349283
Title: A Prospective, Randomized, Double-blind, Parallel-group, Controlled Study of the Immunogenicity and Safety of the Recombinant Hepatitis B Vaccine (Hepavax-Gene TF) and a Comparator Univalent Hepatitis B Vaccine in Neonates
Brief Title: Immunogenicity and Safety of the Hepatitis B Vaccine Hepavax-Gene TF and a Comparator Hepatitis B Vaccine in Newborns
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HVG-V-A002
Record Dates: First submitted 2011-05-05; First posted 2011-05-06 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2013-01

CONDITIONS: Hepatitis B
Keywords: Hepatitis B Vaccine; Hepatitis B Virus; Antigen; Antibody; Vaccination
MeSH Terms: conditions — Hepatitis B | interventions — Engerix-B

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- HepavaxGene Stratum 1a (Experimental): Subjects of mothers with chronic hepatitis B (positive for both HBsAg and hepatitis B envelope antigen - HBeAg)
  Interventions: Biological: HepavaxGene (thiomersal free)
- Comparator vaccine Stratum 1a (Active Comparator): Subjects of mothers with chronic hepatitis B (positive for both HBsAg and HBeAg)
  Interventions: Biological: Engerix B
- HepavaxGene Stratum 1b (Experimental): Subjects of mothers with chronic hepatitis B (positive for HBsAg only)
  Interventions: Biological: HepavaxGene (thiomersal free)
- Comparator vaccine Stratum 1b (Active Comparator): Subjects of mothers with chronic hepatitis B (positive for HBsAg only)
  Interventions: Biological: Engerix B
- HepavaxGene Stratum 2 (Experimental): Subjects of mothers without chronic hepatitis B (negative for both HBsAg and HBeAg)
  Interventions: Biological: HepavaxGene (thiomersal free)
- Comparator vaccine Stratum 2 (Active Comparator): Subjects of mothers without chronic hepatitis B (negative for both HBsAg and HBeAg)
  Interventions: Biological: Engerix B

INTERVENTIONS:
Biological: HepavaxGene (thiomersal free) — 10 µg/0.5 mL, intramuscular injection on Day 1, Month 1, Month 6
  Arms: HepavaxGene Stratum 1a; HepavaxGene Stratum 1b; HepavaxGene Stratum 2
Biological: Engerix B — 10 µg/0.5 mL, intramuscular injection on Day 1, Month 1, Month 6
  Arms: Comparator vaccine Stratum 1a; Comparator vaccine Stratum 1b; Comparator vaccine Stratum 2

SUMMARY:
The primary purpose of this study is to determine whether HepavaxGene TF is non-inferior to the comparator vaccine both at impeding hepatitis B transmission from mothers positive for chronic hepatitis B (Stratum 1) to their children and also in terms of seroconversion rate in children of mothers negative for chronic hepatitis B (Stratum 2) one month after completion of the immunization schedule.

ELIGIBILITY:
Three types of subject:

Neonates whose mothers are positive for both HBsAg and HBeAg

Neonates whose mothers are positive for only HBsAg

Neonates whose mothers are negative for both HBsAg and HBeAg

INCLUSION CRITERIA:

* Full-term neonates with gestational age from 37 weeks to 42 weeks;
* Apgar scores are no less than 7 at birth;
* Neonates with standard body temperature (auxiliary temperature < 37.1°);
* Neonates weighing ≥ 2,500 grams at birth;
* Neonates with icteric index within the normal range (physiologic jaundice is permitted);
* Informed consent form signed by parent/guardian;
* The requirements of the clinical trial protocol can be observed on the basis of the opinion of the investigator.

EXCLUSION CRITERIA:

* Subject's parent has a history of family diseases such as convulsion and brain diseases;
* Mothers have low immunologic function or a history of organ transplantation or hemodialysis;
* Subject's parent is allergic to any composition of Hepatitis B vaccine;
* A family history of thrombocytopenia, or other disturbance of blood coagulation, which may result in a contraindication for intramuscular injection;
* Known immunologic function damage;
* Mothers had received gamma globulin or immunoglobulin injection during pregnancy;
* Any congenital malformation
* Known or suspected to suffer from diseases such as active infection and cardiovascular disease;
* Any condition believed by the investigator to have possible impact on trial evaluation.

Max Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1738 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate for subjects in Stratum 2 | Month 7
  Hepatitis B surface antibody (HBsAb) concentrations are measured from blood samples by standard enzyme linked immuno sorbent assay (ELISA) for subjects whose mothers are negative for chronic hepatitis B. Seroconversion rate is defined as HBsAb ≥10 mIU/mL.
Positivity for HBsAg for subjects in Stratum 1 | Month 2, Month 7 and Month 12
  The presence of hepatitis B surface antigen (HBsAg), as determined by ELISA, for subjects whose mothers are positive for chronic hepatitis B

SECONDARY OUTCOMES:
Seroconversion rate for subjects in Stratum 1 | Month 7
  Seroconversion rate is defined as HBsAb concentrations from ELISA ≥10 mIU/mL
Solicited adverse events | Days 1 to 4
  Local adverse events: pain, erythema, swelling at the injection site Systemic adverse events: irritability, sleepiness, change in eating/breast feeding habits, crying, fever [body temperature ≥38°C]
Seroconversion rate for subjects in Stratum 1 | Month 12
  Seroconversion rate is defined as HBsAb concentrations from ELISA ≥10 mIU/mL
Positivity for HBsAg for subjects in Stratum 2 | Months 2, 7 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Fencai, MD, Principal Investigator — Jiangsu Provincial Center for Disease Prevention and Control, China
Locations (1):
- Center for Disease Control and Prevention Jiangsu Province, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Zhu F, Deckx H, Roten R, Michiels B, Sarnecki M. Comparative Efficacy, Safety and Immunogenicity of Hepavax-Gene TF and Engerix-B Recombinant Hepatitis B Vaccines in Neonates in China. Pediatr Infect Dis J. 2017 Jan;36(1):94-101. doi: 10.1097/INF.0000000000001361. PMID 27753794